CLINICAL TRIAL: NCT06387082
Title: A Multicenter, Open-Label Phase I Clinical Study to Evaluate the Safety, Pharmacokinetics and Efficacy of HMPL-506 in Patients With Hematological Malignancies
Brief Title: A Clinical Study of HMPL-506 in Patients With Hematological Malignancies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hutchmed (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2023-506-00CH1
Record Dates: First submitted 2024-04-19; First posted 2024-04-26 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Hematological Malignancies
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (13):
- 50mg QD (Experimental): The starting dose of 50 mg QD will be escalated using the accelerated titration design in the first enrolled subject.
  If no DLT is observed and no Grade 2 or higher investigational product-related adverse events occur during the DLT observation period at the dose 50mg QD, the dose can be escalated to 100 mg QD, and the mTPI-2 design will be used for dose escalation.
  The dose will be escalated based on available efficacy and safety data in conjunction with preclinical Pharmacodynamics, Pharmacokinetic (PK) and Pharmacodynamics (PD) data.
  Interventions: Drug: HMPL-506
- 100mg QD (Experimental): At least 3 patients will be enrolled at each dose level and additional 3 patients will be recruited at the dose level decided by the next cohort following the rules specified in the protocol when all patients in the current dose group complete the DLT assessment. The number of patients finally enrolled in each dose group is not limited to 3 patients, and the need to increase the number of patients may be decided by the sponsor or by discussion at a SRC meeting to obtain the relevant data required. However, at least 3 DLT evaluable patients per dose group must be ensured.
  Interventions: Drug: HMPL-506
- 200mg QD (Experimental): At least 3 patients will be enrolled at each dose level and additional 3 patients will be recruited at the dose level decided by the next cohort following the rules specified in the protocol when all patients in the current dose group complete the DLT assessment. The number of patients finally enrolled in each dose group is not limited to 3 patients, and the need to increase the number of patients may be decided by the sponsor or by discussion at a SRC meeting to obtain the relevant data required. However, at least 3 DLT evaluable patients per dose group must be ensured.
  Interventions: Drug: HMPL-506
- 300mg QD (Experimental): At least 3 patients will be enrolled at each dose level and additional 3 patients will be recruited at the dose level decided by the next cohort following the rules specified in the protocol when all patients in the current dose group complete the DLT assessment. The number of patients finally enrolled in each dose group is not limited to 3 patients, and the need to increase the number of patients may be decided by the sponsor or by discussion at a SRC meeting to obtain the relevant data required. However, at least 3 DLT evaluable patients per dose group must be ensured.
  Interventions: Drug: HMPL-506
- 400mg QD (Experimental): At least 3 patients will be enrolled at each dose level and additional 3 patients will be recruited at the dose level decided by the next cohort following the rules specified in the protocol when all patients in the current dose group complete the DLT assessment. The number of patients finally enrolled in each dose group is not limited to 3 patients, and the need to increase the number of patients may be decided by the sponsor or by discussion at a SRC meeting to obtain the relevant data required. However, at least 3 DLT evaluable patients per dose group must be ensured.
  Interventions: Drug: HMPL-506
- 25 mg BID (Experimental): At least 3 patients will be enrolled at each dose level and additional 3 patients will be recruited at the dose level decided by the next cohort following the rules specified in the protocol when all patients in the current dose group complete the DLT assessment. The number of patients finally enrolled in each dose group is not limited to 3 patients, and the need to increase the number of patients may be decided by the sponsor or by discussion at a SRC meeting to obtain the relevant data required. However, at least 3 DLT evaluable patients per dose group must be ensured.
  Interventions: Drug: HMPL-506
- 50mg BID (Experimental): At least 3 patients will be enrolled at each dose level and additional 3 patients will be recruited at the dose level decided by the next cohort following the rules specified in the protocol when all patients in the current dose group complete the DLT assessment. The number of patients finally enrolled in each dose group is not limited to 3 patients, and the need to increase the number of patients may be decided by the sponsor or by discussion at a SRC meeting to obtain the relevant data required. However, at least 3 DLT evaluable patients per dose group must be ensured.
  Interventions: Drug: HMPL-506
- 75 mg BID (Experimental): At least 3 patients will be enrolled at each dose level and additional 3 patients will be recruited at the dose level decided by the next cohort following the rules specified in the protocol when all patients in the current dose group complete the DLT assessment. The number of patients finally enrolled in each dose group is not limited to 3 patients, and the need to increase the number of patients may be decided by the sponsor or by discussion at a SRC meeting to obtain the relevant data required. However, at least 3 DLT evaluable patients per dose group must be ensured.
  Interventions: Drug: HMPL-506
- 150mg QD (Experimental): At least 3 patients will be enrolled at each dose level and additional 3 patients will be recruited at the dose level decided by the next cohort following the rules specified in the protocol when all patients in the current dose group complete the DLT assessment. The number of patients finally enrolled in each dose group is not limited to 3 patients, and the need to increase the number of patients may be decided by the sponsor or by discussion at a SRC meeting to obtain the relevant data required. However, at least 3 DLT evaluable patients per dose group must be ensured.
  Interventions: Drug: HMPL-506
- 100mg BID (Experimental): At least 3 patients will be enrolled at each dose level and additional 3 patients will be recruited at the dose level decided by the next cohort following the rules specified in the protocol when all patients in the current dose group complete the DLT assessment. The number of patients finally enrolled in each dose group is not limited to 3 patients, and the need to increase the number of patients may be decided by the sponsor or by discussion at a SRC meeting to obtain the relevant data required. However, at least 3 DLT evaluable patients per dose group must be ensured.
  Interventions: Drug: HMPL-506
- 150mg BID (Experimental): At least 3 patients will be enrolled at each dose level and additional 3 patients will be recruited at the dose level decided by the next cohort following the rules specified in the protocol when all patients in the current dose group complete the DLT assessment. The number of patients finally enrolled in each dose group is not limited to 3 patients, and the need to increase the number of patients may be decided by the sponsor or by discussion at a SRC meeting to obtain the relevant data required. However, at least 3 DLT evaluable patients per dose group must be ensured.
  Interventions: Drug: HMPL-506
- 200mg BID (Experimental): At least 3 patients will be enrolled at each dose level and additional 3 patients will be recruited at the dose level decided by the next cohort following the rules specified in the protocol when all patients in the current dose group complete the DLT assessment. The number of patients finally enrolled in each dose group is not limited to 3 patients, and the need to increase the number of patients may be decided by the sponsor or by discussion at a SRC meeting to obtain the relevant data required. However, at least 3 DLT evaluable patients per dose group must be ensured.
  Interventions: Drug: HMPL-506
- Other dose determined by SRC (Experimental): At least 3 patients will be enrolled at each dose level and additional 3 patients will be recruited at the dose level decided by the next cohort following the rules specified in the protocol when all patients in the current dose group complete the DLT assessment. The number of patients finally enrolled in each dose group is not limited to 3 patients, and the need to increase the number of patients may be decided by the sponsor or by discussion at a SRC meeting to obtain the relevant data required. However, at least 3 DLT evaluable patients per dose group must be ensured.
  Interventions: Drug: HMPL-506

INTERVENTIONS:
Drug: HMPL-506 — HMPL-506 will be administered orally in 28-day cycles, until disease progression/relapse , death, intolerable toxicity, receipt of another anti-tumor therapy (including HSCT), failure to further benefit , patient withdrawal, loss to follow-up or end of the study, whichever comes first.
  Other Names: Two strengths of HMPL-506 tablets (25 mg and 100 mg) will be used for this clinical study

SUMMARY:
This is a Phase 1, multicenter, open-label clinical study of HMPL-506 administered orally in the treatment of hematological malignancies. Only eligible patients who provide the signed informed consent form (ICF) can be enrolled in this study. The study consists of two phases, i.e., a dose escalation phase and a dose expansion phase. The study is expected to enroll approximately 60 to 132 patients, including approximately 30 to 38 patients in the dose escalation phase and approximately 30 to 72 patients in the dose expansion phase.

DETAILED DESCRIPTION:
The study is divided into 2 Phases, Dose Escalation Phase &Dose Expansion Phase.

Dose Escalation Phase: In this phase, the accelerated titration design with the modified toxicity probability interval-2 (mTPI-2) design will be used for dose escalation and determination of the Maximum tolerated dose (MTD). Approximately 30 to 38 patients with MLL-rearranged and/or NPM1-mutant relapsed/refractory Acute Myeloid Leukemia (AML) and Acute Lymphocytic Leukemia (ALL) will be enrolled in this phase.

The determined starting dose of HMPL-506, i.e., 50 mg QD (orally once daily, approximately every 24 hours）, According to the Safety Monitoring Committee (SRC) safety, efficacy and PK/PD data of the first 4 patients in the 50 mg QD dose group of HMPL-506, it was decided to administer the pre dose + therapeutic dose, initially set the pre dose for one week (or duration based on SRC decision), and then continue the treatment at the therapeutic dose.

The Pre-dose is initially set as 25 mg QD (or the lead dose selected according to SRC decision), The preliminary set escalation gradient includes: a. QD dosing: 50 mg, 100 mg, 150 mg, 200 mg, 300 mg, 400 mg, etc.; b. BID dosing: starting dose of 25 mg, 50 mg, 75 mg, 100 mg, 150 mg, 200 mg, etc.; or refer to the SRC-determined incremental gradient.

According to the Safety Monitoring Committee (SRC) safety, efficacy and PK/PD data of the first 4 patients in the 50 mg QD dose group of HMPL-506, it was decided to administer the lead dose + therapeutic dose, initially set the lead dose for one week (or duration based on SRC decision), and then continue the treatment at the therapeutic dose.

The dose will be escalated based on available efficacy and safety data in conjunction with preclinical pharmacodynamics, PK data. safety review committee（SRC） meetings will be held to discuss the necessity of expanding the sample size of 1 or more selected dose groups, with approximately 6 to 10 patients in each dose group, to obtain a sufficient amount of safety and efficacy data.

Dose Expansion Phase: The dose expansion phase will be conducted after the determination of the recommended phase 2 dose(RP2D) and/or Maximum tolerated dose （MTD） and approximately 30 to 60 patients with hematological malignancies will be enrolled to further evaluate the safety, tolerability and preliminary efficacy of HMPL-506. Patients enrolled in this phase will be divided into three cohorts:

* MLL-rearranged and/or NPM1-mutant relapsed/refractory AML
* MLL-rearranged relapsed/refractory ALL
* Relapsed/refractory multiple myeloma (MM), and AML with genetic alterations such as NUP214 or NUP98 fusion

Approximately 10 to 20 patients are planned to be enrolled in each cohort. Enrolled patients will receive oral dose of HMPL-506 at the RP2D in 28-day cycles until disease progression/relapse (except for patients who are assessed by the investigator as continuing receiving benefit from treatment with the investigational product), death, intolerable toxicity, receiving another anti-tumor therapy, failure to further benefit from the treatment as judged by the investigator, patient withdrawal, loss to follow-up or end of the study, whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet all of the following criteria to be eligible for enrolment.

  1. Having understood this study adequately and being voluntary to sign the ICF;
  2. Age ≥18 years;
  3. 1) Dose escalation phase: patient with MLL-rearranged and/or NPM1-mutant relapsed/refractory AML or ALL (confirmed as per the 2022 World Health Organization (WHO) Classification of Myeloid Neoplasms and Acute Leukemia): 2) Dose expansion phase: approximately 10 to 20 patients will be enrolled in each of the following cohorts

     * MLL-rearranged and/or NPM1-mutant relapsed/refractory AML
     * MLL-rearranged relapsed/refractory ALL
     * Relapsed/refractory MM (which can be screened and enrolled without biomarker testing), and AML harboring genetic alterations such as NUP214 or NUP98 fusion
  4. Eastern Cooperative Oncology Group performance status (ECOG PS) of 0 to 2;
  5. Agree to undergo bone marrow aspiration and/or biopsy before and during treatment;
  6. Women patients of childbearing potential must agree to use highly effective contraceptive methods from screening until 30 days after discontinuation of study treatment, and their male partners must use condoms. See Appendix 11 (Definition of Women of Childbearing Potential [WOCBP] and Acceptable and Unacceptable Contraceptive Methods) for more details. And women patients of childbearing potential should agree not to donate eggs (or oocytes) for reproductive purposes during this period.
  7. Male patients with a female partner of childbearing potential must agree to use condoms when having intercourse during the study and within 30 days after discontinuation of the investigational product. Patients should avoid sperm donation or freezing of sperm during the study and within 30 days after discontinuation of the investigational product.

Exclusion Criteria:

* Subjects will be excluded from this study project if they meet any of the following criteria:

  1. Patients who have previously received treatment with menin inhibitors and experienced progression during treatment;
  2. Patients with definite active central nervous system (CNS) leukemia (prior CNS leukemia has been treated and controlled, but a cerebrospinal fluid test through lumbar puncture is required at screening to confirm the absence of CNS involvement);
  3. Serum total bilirubin (TBIL) > 1.5 × the upper limit of normal (ULN), with the exception of the following patients:

     • Patients with Gilbert's disease, with normal alanine aminotransferase (ALT) and aspartate aminotransferase (AST), and serum TBIL ≤ 3 × ULN
  4. ALT or AST > 3 × ULN in the absence of liver involvement with leukemia or ALT or AST > 5 × ULN in the presence of liver involvement with leukemia (the latter criterion is not applicable in the dose escalation phase);
  5. Glomerular filtration rate or creatinine clearance estimated using Cockcroft-Gault formula < 50 mL/min.
  6. International normalized ratio (INR) > 1.5 × ULN or activated partial thromboplastin time (aPTT) > 1.5 × ULN; this criterion is not applicable in patients who are receiving anticoagulant therapy.
  7. Known history of clinically significant liver disease, including viral hepatitis or other types of hepatitis:

     * Patients with hepatitis B (HBV) (HBsAg or HBcAb positive) can be enrolled if they test negative for HBV DNA by PCR, but the HBV DNA test should be performed every cycle
     * Patients with hepatitis C (HCV) can be enrolled if they test negative for HCV RNA by PCR.
  8. Known human immunodeficiency virus (HIV) infection.
  9. Women who are pregnant (with a positive pregnancy test before administration) or breastfeeding.
  10. History of stroke or intracranial hemorrhage within 6 months prior to the first dose of the investigational product.
  11. Patients with other primary malignancies within the last 5 years, but patients with the following non-invasive tumors that have been treated with curative intent are exceptions: basal cell carcinoma of skin, squamous cell carcinoma of skin, in situ carcinoma of cervix and breast cancer in situ.
  12. Patients who meet any of the following cardiac function-related criteria:

      * Any clinically significant abnormal heart rhythm or conduction requiring clinical intervention.
      * Hereditary long QT syndrome or QTcF > 470 msec.
      * Clinically significant cardiovascular diseases, including acute myocardial infarction, unstable angina pectoris, coronary artery bypass grafting within 6 months prior to enrollment, New York Heart Association (NYHA) Class III or above congestive heart failure, left ventricular ejection fraction (LVEF) < 50%, or uncontrolled hypertension (systolic blood pressure > 140 mmHg or diastolic blood pressure > 90 mmHg), or mean heart rate > 100 beats/min on triplicate electrocardiograms (ECGs) at screening.
  13. Receipt of systemic anti-tumor therapy or radiotherapy within 2 weeks prior to initiation of study treatment:

      * For patients with increased peripheral white blood cell count (WBC > 25 × 109/L), use of hydroxycarbamide is allowed to control peripheral WBC before enrollment and during HMPL-506 treatment.
      * Prophylactic intrathecal injection of chemotherapy drugs (cytarabine, dexamethasone and methotrexate) to prevent CNS leukemia is allowed.
  14. Patients who have received HSCT within 60 days before initiation of study treatment, or are receiving immunosuppressive therapy after HSCT at screening, or require medical intervention to control graft versus host disease (GVHD):

      • Patients who use fixed-dose oral glucocorticoids and/or topical glucocorticoids for the treatment of skin GVHD can be enrolled.
  15. Patients who have received treatment with herbal and traditional medicines/their active ingredients with definite anti-tumor activity within 1 week before initiation of study treatment.
  16. Use of potent inducers or inhibitors of CYP3A4 within 2 weeks (3 weeks for St John's wort) or 5 half-lives (whichever is longer) before initiation of study treatment.
  17. An interval of less than 2 weeks from the last dose of any small molecular drug or of less than 4 weeks from the last dose of any macromolecular drug (e.g., antibody drugs) administered during previous participation in other drug clinical trials before treatment initiation in this study.
  18. Patients who have undergone major surgery within 4 weeks prior to the first dose of the investigational product.
  19. Toxicities from previous anti-tumor treatments have not yet recovered to Grade ≤ 1 (excluding alopecia).
  20. Patients with uncontrolled active infection requiring hospitalization or intravenous antibiotics (defined as persistent signs/symptoms related to the infection without improvement despite receipt of appropriate anti-infection therapy and/or other treatments); or unexplained pyrexia with a temperature above 38.5℃ during the screening period (only patients with tumor fever as judged by the investigator can be enrolled);

      • Patients with neutropenia who, in the opinion of the investigator, require prophylactic intravenous antibiotics can be enrolled
  21. Presence of conditions that may affect the absorption of the investigational product as judged by the investigator, such as inability to take drugs orally, past surgery history or severe gastrointestinal diseases including dysphagia and active gastric ulcer.
  22. Patients with poor compliance who are judged by the investigator as not suitable for participation in this clinical study.
  23. Any other disease, metabolic abnormality, physical examination abnormality or clinically significant laboratory test abnormality, based on which the investigator has reason to suspect that the patient has certain disease or condition that is not suitable for treatment with the investigational product, or that will affect the interpretation of study results or will put the patient at high risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2024-05-27 (Actual); Primary Completion 2027-10-08 (Estimated); Study Completion 2027-12-08 (Estimated)

PRIMARY OUTCOMES:
Safety evaluation: Safety Incidence of Dose-limiting Toxicity (DLTs) | The DLT assessment window is Cycle 1 + 3 days (starting from dosing on Day -3, i.e., 28 + 3 days) in the first two dose groups (50 mg and 100 mg), and Cycle 1 (starting from Day 1 of each cycle, i.e., 28 days) in other dose groups.
  Incidence of serious Dose-limiting Toxicity evaluated using the NCI CTCAE V5.0.
Safety evaluation: Incidence of serious adverse events (SAEs) and Relationship to Study Drug | The time from the first dose of HMPL-506 to 30 days after last dose, or initiation of a new anti-tumor therapy, whichever comes first. Maybe assessed up to 42 months
  Incidence of serious adverse events (SAEs) evaluated using the NCI CTCAE V5.0 and the relationship of DLTs and SAEs with the investigational product.
  The assessment window is from the first dose of HMPL-506 to 30 days after last dose, or initiation of a new anti-tumor therapy, whichever comes first.
Efficacy evaluation: Anti-tumor efficacy evaluation. | To assess at every cycle during the first 6 cycles of treatment (each cycle is 28 days) and once every 2 cycles thereafter; response evaluation will also be conducted at each Event-free survival (EFS) follow-up visit.Maybe assessed up to 42 Months.
  Performing anti-tumor efficacy evaluation of HMPL-506 based on Complete response (CR), Complete response with partial recovery of hematology (CRh), Complete response with incomplete hematological recovery (CRi) assessed by the Investigator.
  Response evaluation in AML will be conducted based on the European LeukmiaNet (ELN) 2022 criteria; response evaluation in ALL will be conducted based on the National Comprehensive Cancer Network (NCCN) Guidelines for the Diagnosis and Treatment of ALL (2023 Version 3).

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) and Relationship to Study Drug | The time from the first dose of HMPL-506 to 30 days after last dose, or initiation of a new anti-tumor therapy, whichever comes first. Maybe assessed up to 42 Months.
  Incidence of each type of adverse event evaluated by NCI CTCAE V5.0 and its relationship to study drug
Adverse Events Associated with Dose Modifications | The time from the first dose of HMPL-506 to 30 days after last dose, or initiation of a new anti-tumor therapy, whichever comes first. Maybe assessed up to 42 Months.
  Incidence of adverse events leading to dose interruption, reduction, or treatment discontinuation
Evaluate electrocardiogram (ECG) assessments. | The time from the first dose of HMPL-506 to 30 days after last dose, or initiation of a new anti-tumor therapy, whichever comes first. Maybe assessed up to 42 Months.
  Observe QT interval changes before and after treatment.
Complete response rate (CR rate) | To assess at every cycle during the first 6 cycles of treatment (each cycle is 28 days) and once every 2 cycles thereafter; response evaluation will also be conducted at each EFS follow-up visit.Maybe assessed up to 42 Months.
  Defined as the proportion of subjects achieving CR as assessed by the investigator.Response evaluation in AML will be conducted based on the European LeukmiaNet (ELN) 2022 criteria; response evaluation in ALL will be conducted based on the National Comprehensive Cancer Network (NCCN) Guidelines for the Diagnosis and Treatment of ALL (2023 Version 3).
Complete response (CR)+ Complete response with partial recovery of hematology (CRh) rate | To assess at every cycle during the first 6 cycles of treatment (each cycle is 28 days) and once every 2 cycles thereafter; response evaluation will also be conducted at each EFS follow-up visit.Maybe assessed up to 42 Months.
  Defined as the proportion of subjects achieving CR or CRh as assessed by the investigator. Response evaluation in AML will be conducted based on the European LeukmiaNet (ELN) 2022 criteria; response evaluation in ALL will be conducted based on the National Comprehensive Cancer Network (NCCN) Guidelines for the Diagnosis and Treatment of ALL (2023 Version 3)
Composite complete response (CRc) rate | To assess at every cycle during the first 6 cycles of treatment (each cycle is 28 days) and once every 2 cycles thereafter; response evaluation will also be conducted at each EFS follow-up visit.Maybe assessed up to 42 Months.
  Defined as the proportion of subjects achieving CR, CRh, or CRi(incomplete hematological recovery) as assessed by the investigator.
  Response evaluation in AML will be conducted based on the European LeukmiaNet (ELN) 2022 criteria; response evaluation in ALL will be conducted based on the National Comprehensive Cancer Network (NCCN) Guidelines for the Diagnosis and Treatment of ALL (2023 Version 3)
Objective response rate (ORR) | To assess at every cycle during the first 6 cycles of treatment (each cycle is 28 days) and once every 2 cycles thereafter; response evaluation will also be conducted at each EFS follow-up visit.Maybe assessed up to 42 Months.
  defined as the proportion of patients with CR, CRh, CRi, morphologic leukemia-free status (MLFS), and partial response (PR) as judged by the investigator.
  Response evaluation in AML will be conducted based on the European LeukmiaNet (ELN) 2022 criteria; response evaluation in ALL will be conducted based on the National Comprehensive Cancer Network (NCCN) Guidelines for the Diagnosis and Treatment of ALL (2023 Version 3)
Time to Complete response (CR)+Complete response with partial recovery of hematology (CRh) | To assess at every cycle during the first 6 cycles of treatment (each cycle is 28 days) and once every 2 cycles thereafter; response evaluation will also be conducted at each EFS follow-up visit.Maybe assessed up to 42 Months.
  Defined as the time from the first administration of HMPL-506 to the first occurrence of CR/CRh.
  Response evaluation in AML will be conducted based on the European LeukmiaNet (ELN) 2022 criteria; response evaluation in ALL will be conducted based on the National Comprehensive Cancer Network (NCCN) Guidelines for the Diagnosis and Treatment of ALL (2023 Version 3)
Time to Complete response (CR)+Complete response with partial recovery of hematology (CRh) +incomplete hematological recovery (CRi) | To assess at every cycle during the first 6 cycles of treatment (each cycle is 28 days) and once every 2 cycles thereafter; response evaluation will also be conducted at each EFS follow-up visit.Maybe assessed up to 42 Months.
  Defined as the time from the first administration of HMPL-506 to the first occurrence of CR/CRh/CRi.
  Response evaluation in AML will be conducted based on the European LeukmiaNet (ELN) 2022 criteria; response evaluation in ALL will be conducted based on the National Comprehensive Cancer Network (NCCN) Guidelines for the Diagnosis and Treatment of ALL (2023 Version 3)
Time to disease response (TTR) | To assess at every cycle during the first 6 cycles of treatment (each cycle is 28 days) and once every 2 cycles thereafter; response evaluation will also be conducted at each EFS follow-up visit.Maybe assessed up to 42 Months.
  Defined as the time from the first administration of HMPL-506 to the first achievement of CR/CRh/CRi/MLFS/PR.
  Response evaluation in AML will be conducted based on the European LeukmiaNet (ELN) 2022 criteria; response evaluation in ALL will be conducted based on the National Comprehensive Cancer Network (NCCN) Guidelines for the Diagnosis and Treatment of ALL (2023 Version 3)
Duration of Complete response (CR)+Complete response with partial recovery of hematology (CRh) | To assess at every cycle during the first 6 cycles of treatment (each cycle is 28 days) and once every 2 cycles thereafter; response evaluation will also be conducted at each EFS follow-up visit.Maybe assessed up to 42 Months.
  Defined as the time from first achievement of CR/CRh until disease recurrence, progression, or death from any cause, whichever occurs first.
  Response evaluation in AML will be conducted based on the European LeukmiaNet (ELN) 2022 criteria; response evaluation in ALL will be conducted based on the National Comprehensive Cancer Network (NCCN) Guidelines for the Diagnosis and Treatment of ALL (2023 Version 3)
Duration of response (DOR) | To assess at every cycle during the first 6 cycles of treatment (each cycle is 28 days) and once every 2 cycles thereafter; response evaluation will also be conducted at each EFS follow-up visit.Maybe assessed up to 42 Months.
  Defined as the time from the patient 's first achievement of CR/CRh/CRi/MLFS/PR until disease recurrence, progression, or death from any cause, whichever came first.
  Response evaluation in AML will be conducted based on the European LeukmiaNet (ELN) 2022 criteria; response evaluation in ALL will be conducted based on the National Comprehensive Cancer Network (NCCN) Guidelines for the Diagnosis and Treatment of ALL (2023 Version 3).
Event-free survival (EFS) | To assess at every cycle during the first 6 cycles of treatment (each cycle is 28 days) and once every 2 cycles thereafter; response evaluation will also be conducted at each EFS follow-up visit.Maybe assessed up to 42 Months.
  Defined as the time from the start of treatment to the date of loss of response, hematologic relapse after CR/CRh/CRi, or death from any cause, whichever came first.
  Response evaluation in AML will be conducted based on the European LeukmiaNet (ELN) 2022 criteria; response evaluation in ALL will be conducted based on the National Comprehensive Cancer Network (NCCN) Guidelines for the Diagnosis and Treatment of ALL (2023 Version 3).
Relapse-free survival (RFS) | To assess at every cycle during the first 6 cycles of treatment (each cycle is 28 days) and once every 2 cycles thereafter; response evaluation will also be conducted at each EFS follow-up visit.Maybe assessed up to 42 Months.
  (For patients who achieved CR/CRh/CRi only) Defined as the time from achievement of response (CR/CRh/CRi) to hematologic relapse, death from any cause, whichever came first. hematologic relapse after CR/CRh/CRi, or death from any cause, whichever came first.
  Response evaluation in AML will be conducted based on the European LeukmiaNet (ELN) 2022 criteria; response evaluation in ALL will be conducted based on the National Comprehensive Cancer Network (NCCN) Guidelines for the Diagnosis and Treatment of ALL (2023 Version 3).
Overall survival (OS) | Until to disease progression/relapse or initiate new anti-tumor therapies will continue to attend OS follow-up visits every 2 months until death, patient withdrawal, loss to follow-up or end of study, whichever comes first, Maybe assessed up to 42 Months
  Defined as the time from the start of study drug until death from any cause. Response evaluation in AML will be conducted based on the European LeukmiaNet (ELN) 2022 criteria; response evaluation in ALL will be conducted based on the National Comprehensive Cancer Network (NCCN) Guidelines for the Diagnosis and Treatment of ALL (2023 Version 3).
Pharmacokinetic analysis-Maximum concentration (Cmax) | The window is before the first dose of HMPL-506 to Cycle 3 Day1(each cycle is 28 days).
  To characterized Maximum concentration (Cmax) of HMPL-506 and metabolite M7 in plasma and bone marrow were measured before and after treatment.
Pharmacokinetic analysis: Peak time (Tmax) | The access window is before the first dose of HMPL-506 to Cycle 3 Day1(each cycle is 28 days).12 Weeks.
  To characterized Peak time (Tmax)of HMPL-506 and metabolite M7 in plasma and bone marrow were measured before and after treatment.
Pharmacokinetic analysis: Clearance half-life (T1/2) | The access window is before the first dose of HMPL-506 to Cycle 3 Day1(each cycle is 28 days).12 Weeks.
  To characterized Clearance half-life (T1/2) of HMPL-506 and metabolite M7 in plasma and bone marrow were measured before and after treatment.
Pharmacokinetic analysis: area under the plasma concentration-time curve (AUC0-t) | The access window is before the first dose of HMPL-506 to Cycle 3 Day1(each cycle is 28 days).12 Weeks.
  To characterized area under the plasma concentration-time curve (AUC0-t) of HMPL-506 and metabolite M7 in plasma and bone marrow were measured before and after treatment.

OTHER OUTCOMES:
Evaluate the changes of the Pharmacodynamic Biomarker | the time before the first dose of HMPL-506 to 30 days after last dose or Disease progression.Maybe assessed up to 42 Months.
  Changes in Pharmacodynamic biomarkers (e.g., MEIS3, HOXA9, CD11b etc.) before and after HMPL506 administration, and correlations with dosing and efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Jianxiang Wang, Master, Principal Investigator — Blood Diseases Hospital, Chinese Academy of medical Sciences; Hui Wei, Master, Principal Investigator — Blood Diseases Hospital, Chinese Academy of medical Sciences
Locations (16):
- China (16):
  - Xiangya Hospital of Central South University, Changsha
  - First Affiliated Hospital of Chongqing Medical University, Chongqing
  - Fujian Medical University Union Hospital, Fuzhou
  - Nanfang Hospital, Southern Medical University, Guangzhou
  - Sun Yat-sen University Cancer Center, Guangzhou
  - The Affiliated Hospital of Guizhou Medical University, Guiyang
  - The First Affiliated Hospital, Zhejiang University, Hangzhou
  - Anhui Provincial Hospital, Hefei
  - Qilu Hospital of Shandong University, Jinan
  - The First Affiliated Hospital with Nanjing Medical University, Nanjing
  - Shengjing Hospital of China Medical University, Shenyang
  - The First Affiliated Hospital of Soochow University, Suzhou
  - Blood Diseases Hospital, Chinese Academy of medical Sciences, Tianjin
  - Tianjin People's Hospital, Tianjin
  - Wuhan Union Hospital of China, Wuhan
  - Henan Cancer Hospital, Zhengzhou

IPD SHARING:
Plan to Share IPD: No